CLINICAL TRIAL: NCT00456755
Title: A Herbal Formula (SBL) for the Treatment of Perennial Allergic Rhinitis: A Randomized, Double-blind, Placebo-controlled Clinical Trial
Brief Title: Herbal Treatment for Perennial Allergic Rhinitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Zhao Yu, Department of Otorhinolaryngology, Head & Neck Surgery, West China Hospital, Sichuan University, Institute of Chinese Medicine, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ICM/CTS/03/333
Record Dates: First submitted 2007-04-04; First posted 2007-04-05 (Estimated); Results first posted 2010-01-06 (Estimated); Last update posted 2010-01-06 (Estimated); Status verified 2009-11

CONDITIONS: Perennial Allergic Rhinitis
Keywords: Perennial Allergic rhinitis; Traditional Chinese Medicine
MeSH Terms: conditions — Rhinitis, Allergic, Perennial | interventions — Shi-Bi-Lin herbal formula

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Shi-Bi-Lin (Active Comparator): Consist of 6 herbal. 7.5 g Xanthium sibiricum Patrin ex Widder (Asteraceae, Fructus), 20 g Angelica dahurica (Fisch. ex Hoffm.) Benth. (Apiaceae, Radix), 7.5 g Saposhnikovia divaricata (Turcz.) Schischk. (Apiaceae, Radix),15 g Magnolia biondii Pamp., (Magnoliaceae, Flos), 5 g Gentiana scabra Bunge (Gentianaceae, Radix) and 5 g Verbena officinalis L. (Verbenaceae, Herba).
  Interventions: Drug: Shi-Bi-Lin
- Placebo (Placebo Comparator): The placebo contained brown colored starch resembling the SBL powder
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Shi-Bi-Lin — 4 weeks of treatment, dose of 1 g (two capsules), twice daily
  Other Names: Modified from the classic formula Cang-Er-Zi-San.
  Arms: Shi-Bi-Lin
Other: Placebo — 4 weeks of colormatched placebo capsules, dose of 1 g (two capsules), twice daily
  Arms: Placebo

SUMMARY:
Allergic rhinitis(AR) is one of the most common allergic disorders throughout the world.The conventional therapies are effective in alleviating symptoms but the efficacy are limited and not persistent. Furthermonre, the cost and side-effect are known defects. A classical Chinese herbal formula, has been used for AR for centries. Our study purpose is to evaluate the clinical efficacy and safety of this formula verus placebo in perennial allergic rhinitis (PAR).

Hypothesis: the classical herbal formula would improve the symptoms of PAR patients and change some immunological parameters in the peripheral blood when comparing with the placebo.

DETAILED DESCRIPTION:
It is a randomized, double-blind, placebo-controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 18 to 65 years old
* Have typical symotoms of PAR including rhinirrhea, sneezing, nasal obstruction and itching in nose and eyes for at least 2 previous consecutive years.
* Postive skin prick test(SPT) to hose dust mite, mold, animal dander and cockcroach with regular AR medications withould for 3 days prior to the test

Exclusion Criteria:

* Pregnant women and women at risk of conception
* Received allergen injections in previous 2 years
* Regular medications for AR or cold and other allergic disorder
* Seasonal allergic rhinitis, vasomotor rhinitis and rhinitis medicamentosa
* Nasal structure deformities, nasal polyps and hypertrophic rhinitis
* Systematic cortisosteroid used within recent 3 months or nasal cortisosteroid with 15 days
* Other active respiratory disorders
* Active medical disorders: cancer, infection, hematology, renal, hepatic, cardiovascular, metabolic and gastrointestinal diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2004-03; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhao Yu, PhD, Principal Investigator — Department of ENT, Prince of Wales Hospital, The Chinese University of Hong Kong
Locations (2):
- Hong Kong (2):
  - Department of ENT, Prince of Wales Hospital, Hong Kong
  - Department of ENT, Yan Chai Hospital, Hong Kong

REFERENCES:
- [Background] Leung R, Ho P. Asthma, allergy, and atopy in three south-east Asian populations. Thorax. 1994 Dec;49(12):1205-10. doi: 10.1136/thx.49.12.1205. PMID 7878553
- [Background] Spector SL. Overview of comorbid associations of allergic rhinitis. J Allergy Clin Immunol. 1997 Feb;99(2):S773-80. doi: 10.1016/s0091-6749(97)70126-x. PMID 9042070
- [Background] Worldwide variation in prevalence of symptoms of asthma, allergic rhinoconjunctivitis, and atopic eczema: ISAAC. The International Study of Asthma and Allergies in Childhood (ISAAC) Steering Committee. Lancet. 1998 Apr 25;351(9111):1225-32. PMID 9643741
- [Background] Nash DB, Sullivan SD, Mackowiak J. Optimizing quality of care and cost effectiveness in treating allergic rhinitis in a managed care setting. Am J Manag Care. 2000 Jan;6(1 Suppl):S3-15; quiz S19-20. PMID 11009751
- [Background] Bielory L, Lupoli K. Herbal interventions in asthma and allergy. J Asthma. 1999;36(1):1-65. doi: 10.3109/02770909909065150. PMID 10077136
- [Background] Ziment I, Tashkin DP. Alternative medicine for allergy and asthma. J Allergy Clin Immunol. 2000 Oct;106(4):603-14. doi: 10.1067/mai.2000.109432. PMID 11031328
- [Background] Schmolz M, Ottendorfer D, Marz RW, Sieder C. Enhanced resistance to Sendai virus infection in DBA/2J mice with a botanical drug combination (Sinupret). Int Immunopharmacol. 2001 Sep;1(9-10):1841-8. doi: 10.1016/s1567-5769(01)00108-4. PMID 11562075

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started at Jan 2004. Patients were recruited as volunteers from the Prince of Wales hospital, the Yan Chai hospital and the Alice Ho Mui Ling Nethersole Hospital specialist clinics.
Pre-assignment Details: Confirmed perennial allergic rhinitis and have a positive skin test to house-dust mite, mold antigens and/or animal dander was required. Enter 1-week run-in-period, during which symptom diary was given to each subject for the evaluation of symptoms. Eligible case with total score higher than 4.
Period: Overall Study
Arm/Group | Shi-Bi-Lin | Placebo
Started | 63 | 63
Completed | 61 | 62
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Shi-Bi-Lin | Placebo | Total
Number analyzed (Participants) | 63 | 63 | 126
Age Continuous [Mean (Standard Deviation); unit: Year]
  Age | 41.19 (12.38) | 36.02 (11.14) | 38.60 (12.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 43 | 83
  Male | 23 | 20 | 43
Region of Enrollment [Number; unit: participants]
  Hong Kong | 63 | 63 | 126

OUTCOME MEASURES:

1. Primary Outcome: Allergic Rhinitis Symptom Score Including Rhinorrhea, Nasal Obstruction, Sneezing, Itchy Nose and Itchy Eyes at Week 4
Description: The severity of PAR was evaluated by means of a daily symptom diary chart. Patients were instructed to grade retrospectively everyday before bedtime, their generalwell-being, nasalsymptoms (nasal blockage, rhinorrhea, nose itching, sneezing) and non-nasal symptoms(itching eyes, tearing eyes, redness of eyes, itching of ears or palate) on the diary chart. A 4-point severity scale from no symptoms (0), mild (1), moderated (2) to severe (3) was used.
Time Frame: 4 week
Measure: Mean (Standard Deviation); unit: Unit Score
Arm/Group | Shi-Bi-Lin | Placebo
Number analyzed (Participants) | 63 | 63
Unit Score
  General Health | 2.82 (0.8) | 2.8 (0.78)
  Nose Blockage | 1.19 (0.68) | 1.21 (0.77)
  Rhinorrhea volume | 1.26 (0.71) | 1.24 (0.7)
  Sneeze Frequency | 1.15 (0.64) | 1.18 (0.70)
  Nose Itching | 1.11 (0.58) | 0.99 (0.75)
  Eyes Itching | 0.73 (0.67) | 0.56 (0.76)
  Tears | 0.52 (0.71) | 0.43 (0.67)
  Eye Congestion | 0.37 (0.6) | 0.26 (0.58)
  Ear itching | 0.81 (0.65) | 0.61 (0.78)

2. Secondary Outcome: Quality of Life (Difference Between Baseline and Week 4)
Description: SF-36 QOL questionnaire administrated before and after treatment. It has eight domains: general health (GH), physical functioning (PF), social functioning (SF), role limitation caused by physical problems (RP), bodily pain (BP), role limitations caused by emotional problem (RE), mental health (MH), and vitality (VT). Each domain was started from 0 (worst health) to 100 (best health).
Time Frame: 4 week
Population: ITT
Measure: Mean (Standard Deviation); unit: Unit Score
Arm/Group | Shi-Bi-Lin | Placebo
Number analyzed (Participants) | 63 | 63
Unit Score
  Physical functioning | 4 (14) | 0 (10)
  Role limitation by physical problem | 7 (33) | 3 (30)
  Bodily pain | -3 (25) | -10 (21)
  General Health | -7 (20) | -9 (23)
  Vitality | 8 (22) | 13 (20)
  Socail functioning | 17 (18) | 17 (19)
  Role limitation by emotional problem | 13 (29) | 3 (28)
  Mental health | 1 (23) | 1 (18)

ADVERSE EVENTS:
Time Frame: During the 4 week Follow up visit, clients may report any Adverse Event they experience.
Arm/Group | Shi-Bi-Lin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/63
Other Adverse Events (participants affected / at risk) | 0/63 | 0/63

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No